CLINICAL TRIAL: NCT01504763
Title: Measuring the Effect of Chair Massage on Stress Related Symptoms for Nurses: A Pilot Study
Brief Title: Measuring the Effect of Chair Massage on Stress Related Symptoms for Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deborah Engen, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08-004874
Record Dates: First submitted 2011-12-21; First posted 2012-01-05 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Stress; Fatigue; Anxiety; Tension
Keywords: Massage; Chair massage; Relaxation; Nurses
MeSH Terms: conditions — Fatigue; Anxiety Disorders | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Massage (Experimental): Chair massage for 15 minutes once a week for 10 weeks.
  Interventions: Procedure: Chair massage

INTERVENTIONS:
Procedure: Chair massage — Chair massage for 15 minutes once a week for 10 weeks.
  Other Names: Massage

SUMMARY:
The purpose of this study was to assess the feasibility and effect of chair massage provided during working hours for nurses in an inpatient psychiatric and an outpatient pain rehabilitation unit and on the nurses stress related symptoms.

DETAILED DESCRIPTION:
Nursing staff working in a hospital in-patient psychiatric unit and out-patient pain rehabilitation/ fibromyalgia units each have varying causes of stress as both are intensely demanding environments. The physical and psychosocial demands of these stress-loaded work environments place a significant amount of strain on the physiological well-being of the employee.

Nurses in these settings are considered healthy employees and able to participate in the workforce, although symptoms such as headaches, shoulder tension, insomnia, fatigue, and muscle and joint pain are often a part of their work day. As these stress related symptoms become more chronic, they lead to days missed and become pre-cursors to physiological illnesses so warrant further search for prevention tactics.

Massage therapy has been noted to decrease levels of anxiety and fatigue which is essential to maintaining employee's efficient care in a dynamic environment. This study will provide massage in the workplace utilizing chair massage as it is easy to set up, does not need a great deal of space, and can be provided in semi-private areas, as the participant remains clothed. A 2006 report on a small study indicated chair massage can be effective in reducing stress perception in nurses within a hospital setting, at least in the short-term. Another study reported some short-term positive effects on stress related symptoms; and came to the conclusion that further studies are indicated to examine the efficacy of workplace-based massage therapy programs.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-65 able to give informed consent
* Able to speak and understand English
* Minimum of 8-hour per day shift schedule with .75 - 1.0 FTE.
* Need to be able to schedule one massage per week in the available massage schedule time slots.

Exclusion Criteria:

* Individuals being treated for acute musculoskeletal symptoms
* Individuals currently on work restrictions
* Undergoing treatments for a malignancy
* Pregnancy (due to this being chair massage)
* Recent head, neck, shoulder or back surgeries
* Pins or joint fusion of the head or neck
* Current sinus infections, earaches, or vascular migraines
* Nursing staff that float on to the unit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in stress, anxiety and quality of life after 10 weeks of chair massage therapy in nursing staff using four self reported instruments. | 10 Weeks

SECONDARY OUTCOMES:
Change from baseline of stress related symptoms in nursing staff at 5 weeks. | 5 Weeks
Change from baseline of stress related symptoms in nursing staff at 10 weeks. | 10 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J. Engen, O.T., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States